CLINICAL TRIAL: NCT05343364
Title: A Phase 1, Randomized, Parallel-group, Open-label, Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Vonoprazan (10 or 20 mg Once Daily) in Adolescents With Symptomatic Gastroesophageal Reflux Disease
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Vonoprazan in Adolescents With Symptomatic Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VPED-102
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Vonoprazan; Gastroesophageal Reflux; GERD; Adolescents; Pharmacokinetics
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 10 mg (Experimental): Participants will receive vonoprazan 10 mg once daily for 14 days.
  Interventions: Drug: Vonoprazan
- Vonoprazan 20 mg (Experimental): Participants will receive vonoprazan 20 mg once daily for 14 days.
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Oral Tablet

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic profile of vonoprazan in adolescent participants with symptomatic gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* The participant is 12 to 17 years of age, inclusive, at the time of informed consent signing and throughout study participation.
* The participant has a body weight within the 5th through 95th percentile by age, inclusive, as determined by the National Center for Health Statistics.
* The participant has a medical history of symptoms of GERD for at least 3 months prior to screening, based on physical examination, current symptoms (eg, heartburn), or diagnostic tests (eg, pH or endoscopy). Notes in the medical records and/or other source documents such as prior endoscopies can be used to support the diagnosis.
* The participant has symptoms of at least moderate heartburn severity based on the GERD Symptom Assessment-Investigator scale performed at screening.
* The participant must be able to swallow study drug.
* Parent or legal guardian (ie, legally authorized representative [LAR]) is willing and able to complete the informed consent process and comply with study procedures and visit schedule. The participant will provide assent as applicable.
* A female participant of childbearing potential who is or may be sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until 2 weeks after the last dose of study drug.

Exclusion Criteria:

* The participant has used prescription or non-prescription proton pump inhibitors (PPIs) or histamine-2 receptor antagonists (H2RAs) within 7 days prior to randomization or requires their use during the Treatment Period.
* The participant has used sucralfate or antacids within 1 day prior to randomization or requires their use during the Treatment Period.
* The participant has received other agents affecting digestive organs, including muscarinic antagonists (eg, hyoscyamine), prokinetics, oral anticholinergic agents, prostaglandins, bismuth from 30 days prior to Day 1 or requires their use during the course of the study.
* The participant has received atazanavir sulfate or rilpivirine hydrochloride from 5 days prior to Day 1 or requires their use during the course of the study.
* The participant has received any investigational compound (including vonoprazan) within 30 days prior to the start of the Screening Period.
* The participant is an immediate family member or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, child, sibling) or who may have consented under duress.
* The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Period.
* The participant has undergone prior gastrointestinal surgeries such as fundoplication.
* The participant has any abnormal laboratory test values at the start of the Screening Period.
* The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, and titanium oxide, or red or yellow ferric oxide).
* The participant used any prescription (excluding hormonal birth control) or over-the-counter medications (including CYP3A4 inducers), including herbal or nutritional supplements, within 14 days (or 5 half-lives) before the first dose of study drug or throughout the study. NOTE: Acid suppressive therapies are considered separately under exclusion criteria 1 and 2.
* The participant has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or other food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days (or 5 half-lives) before the first dose of study drug or throughout the study.
* Female participant has a positive pregnancy test at screening or check in or is lactating.
* The participant has a positive urine drug or alcohol result at screening.
* The participant has positive results at screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus.
* In the opinion of the investigator, the participant is not suitable for entry into the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (10):
- United States (10):
  - University of South Alabama (USA) Physicians Group, Mobile, Alabama
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Advanced Research Center - Elligo, Anaheim, California
  - Infinite Clinical Trials, Morrow, Georgia
  - Legacy Clinical Solutions: Tandem Clinical Research, LLC, Marrero, Louisiana
  - Boston Specialists, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - PriMED Clinical Research, Dayton, Ohio
  - ARC Clinical Research at Four Points, Austin, Texas
  - Pediatric Gastro, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants were enrolled into this study in the United States between May 2022 and June 2023.
Pre-assignment Details: The total duration of the study was up to 8 weeks. The Screening Period was up to 4 weeks, Treatment Period was 2 weeks, and safety follow-up phone call was 2 weeks after last study drug administration.
Groups:
- Vonoprazan 10 mg QD: Participants were randomized to receive vonoprazan 10 mg once daily (QD) from Day 1 to Day 14.
- Vonoprazan 20 mg QD: Participants were randomized to receive vonoprazan 20 mg QD from Day 1 to Day 14.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: inclusive of all participants who received at least 1 dose of study drug.
Groups:
- Vonoprazan 10 mg QD: Participants were randomized to receive vonoprazan 10 mg QD from Day 1 to Day 14.
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.78) | 15.2 (1.75) | 14.8 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Drug Concentration at Steady State (Cmax-ss) of Vonoprazan
Description: Plasma pharmacokinetic (PK) parameters were estimated using a non-linear mixed effects model and were determined from the concentration-time data for all evaluable participants. Actual sampling times, rather than scheduled or nominal sampling times, were used in all computations using sampling time.
Time Frame: Blood samples were collected predose, once between 0.5 and 2 hours, and once between 2.5 and 4 hours post-dose on Days 7 and 14
Population: PK set: inclusive of all evaluable participants who had at least one measurable concentration result.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Number analyzed (Participants) | 9 | 8
ng/mL | 13.4 [6.57 to 25.6] | 26.7 [13.1 to 49.1]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Interval τ (AUCτ) of Vonoprazan
Description: PK parameters were estimated using a non-linear mixed effects model and were determined from the concentration-time data for all evaluable participants. Actual sampling times, rather than scheduled or nominal sampling times, were used in all computations using sampling time.
Time Frame: as for outcome 1
Population: PK set: inclusive of all evaluable participants who had at least one measurable concentration result.
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Number analyzed (Participants) | 9 | 8
h*ng/mL | 94.6 [56.0 to 165] | 208 [95.6 to 381]

3. Primary Outcome: Apparent Oral Clearance (CL/F) of Vonoprazan
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK set: inclusive of all evaluable participants who had at least one measurable concentration result.
Measure: Mean (Full Range); unit: L/h
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Number analyzed (Participants) | 9 | 8
L/h | 124 [60.5 to 179] | 117 [52.5 to 209]

4. Primary Outcome: Apparent Central Volume of Distribution (Vc/F) of Vonoprazan
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK set: inclusive of all evaluable participants who had at least one measurable concentration result.
Measure: Mean (Full Range); unit: liters
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Number analyzed (Participants) | 9 | 8
liters | 686 [314 to 1280] | 704 [311 to 1110]

5. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: AE: any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug.
  Treatment-emergent adverse event (TEAE): any AE that occurred after the first dose of study drug or at baseline that worsens in either intensity or frequency after the first dose of study drug.
  Serious AE: any AE for which the following occurred: death, was life threatening, hopsitalization or prolongation of hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, or the AE was deemed an important medical event.
  Related AE: any AE that follows a reasonable temporal sequence from administration of study drug, or for which possible involvement of the drug cannot be ruled out, although factors other than the study drug may also be responsible.
  Clinically significant changes from baseline in laboratory test values, (hematology, serum chemistry and urinalysis), electrocardiograms and vital signs were reported as AEs.
Time Frame: Up to Day 28
Population: Safety Set: inclusive of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
Number analyzed (Participants) | 12 | 12
Participants
  Any TEAEs | 4 | 1
  Any Serious TEAEs | 0 | 0
  Any Study Drug-related TEAEs | 0 | 0
  Any Serious Study Drug-related TEAEs | 0 | 0
  Any TEAE Leading to Treatment Discontinuation | 0 | 0
  Any TEAE Leading to Study Discontinuation | 0 | 0
  Any AEs Leading to Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety Set: inclusive of all participants who received at least 1 dose of study drug.
Arm/Group | Vonoprazan 10 mg QD | Vonoprazan 20 mg QD
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg QD (N=12) | Vonoprazan 20 mg QD (N=12)
Cellulitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) are not permitted to publish the data. Data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the PIs to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority over all such issues.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT05343364/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT05343364/SAP_001.pdf